CLINICAL TRIAL: NCT05018598
Title: A 26 Week, Randomized, Double Blind, Multinational, Multicenter, Active Controlled, 2-arm Parallel Group Trial Comparing CHF 5993 100/6/12.5 μg pMDI (Fixed Combination of Extrafine Formulation of Beclometasone Dipropionate Plus Formoterol Fumarate Plus Glycopyrronium Bromide) to CHF 1535 200/6 μg pMDI (Fixed Combination of Extrafine Formulation of Beclometasone Dipropionate Plus Formoterol Fumarate) in Subjects With Asthma Uncontrolled on Medium Doses of Inhaled Corticosteroids in Combination With Long-Acting β2-Agonists.
Brief Title: Step-up to Medium Strength Triple Therapy vs High Strength ICS/LABA in Adult Asthmatics Uncontrolled on Medium Strength ICS/LABA
Acronym: MiSTIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was prematurely stopped due to extensive challenges in patient recruitment. The Sponsor issued a notification of early study termination to all investigational sites and all external stakeholders.
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993AB1-06; 2021-002391-39 (EudraCT Number)
Record Dates: First submitted 2021-08-02; First posted 2021-08-24 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The extension phase will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF5993 100/6/12.5 μg (main phase and extension phase) (Experimental): Main phase: 2 inhalations BID, Daily dose is 400/24/50 μg x 26 weeks
  Open-label extension phase: 2 inhalations BID, Daily dose is 400/24/50 μg x 24 weeks
  Interventions: Drug: Administration via pressurized metered dose inhaler (pMDI)
- CHF1535 200/6 μg (main phase) / CHF5993 200/6/12.5 μg (extension phase only) (Active Comparator): Main phase: 2 inhalations BID, Daily dose is 800/24 μg x 26 weeks
  Open-label extension phase: 2 inhalations BID, Daily dose is 800/24/50 μg x 24 weeks
  Interventions: Drug: Administration via pressurized metered dose inhaler (pMDI)

INTERVENTIONS:
Drug: Administration via pressurized metered dose inhaler (pMDI) — CHF5993 pMDI
  Arms: CHF5993 100/6/12.5 μg (main phase and extension phase)
Drug: Administration via pressurized metered dose inhaler (pMDI) — CHF1535 pMDI or CHF5993 pMDI
  Arms: CHF1535 200/6 μg (main phase) / CHF5993 200/6/12.5 μg (extension phase only)

SUMMARY:
The purpose of this phase IV Study is to compare the efficacy of CHF5993 (BDP/FF/GB 100/6/12.5 pMDI) on uncontrolled asthma subjects, versus CHF1535 (BDP/FF 200/6 pMDI).

The open label extension part aims to assess the proportion of subjects whose asthma remains or becomes adequately controlled..

DETAILED DESCRIPTION:
The study consists in two phases:

The study population includes 1400 subjects that are randomly assigned to two treatment arms. Each participant will be followed for 26 weeks to assess the efficacy of CHF5993 (BDP/FF/GB 100/6/12.5 pMDI).

The study population of the extension part includes 800 subjects who opt to enroll into this extension and receive either CHF5993 (BDP/FF/GB 100/6/12.5 pMDI) or CHF5993 (BDP/FF/GB 200/6/12.5 pMDI) depending on their asthma control status at the end of the main phase.

ELIGIBILITY:
Main phase:

Inclusion Criteria:

1. Informed consent: Subject's written informed consent obtained prior to any study related procedures;
2. Sex and age: Male or female subjects aged ≥ 18 and ≤ 75 years;
3. Diagnosis of asthma: A documented diagnosis of persistant asthma for at least 1 year according to GINA recommendations (Box 1-2, GINA report 2021), and with diagnosis before the subject's age of 40 years;
4. Stable asthma therapy: a stable treatment with medium dose of Inhaled corticosteroids (ICS) (extrafine BDP daily dose > 200 and ≤400 µg or estimated clinically comparable dose, as described in GINA 2021 box 3-6) plus a long-acting ß2-agonist (LABA) (formoterol 24 µg or salmeterol 100 µg or vilanterol 25 µg or other approved dose of LABA as clinically comparable to the others) for at least 4 weeks prior to screening;
5. Lung function: A pre bronchodilator FEV1 < 80% of the predicted normal value, after appropriate washout from bronchodilators, at the screening and randomization visits;
6. Bronchodilator responsiveness: A demonstrated increase in FEV1 > 12% and > 200 mL over baseline within 30 minutes after inhaling 400 µg of salbutamol pMDI (based on ATS/ERS guidelines);
7. A Post-bronchodilator FEV1/FVC ratio ≥ 0.5 within 30 minutes after inhaling 400 µg of salbutamol pMDI at screening (based on ATS/ERS guidelines);
8. Poor Asthma control: Evidence of poorly controlled or uncontrolled asthma as based on an Asthma Control Questionnaire© (ACQ-7) score ≥ 1.5 at screening and at randomization;
9. History of asthma exacerbations: A documented history of one or more asthma exacerbations requiring treatment with systemic corticosteroids or emergency department visit or inpatient hospitalization in the last 3 years prior to screening;
10. A willingness and ability:

    * to correctly use the pMDI inhalers;
    * to perform all trial related procedures including technically acceptable pulmonary function tests;
    * to correctly use the e-Diary/e-Peak flow meter.
11. Female subjects:

    a. Woman of Childbearing Potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up call or ii. WOCBP with non-fertile male partners (contraception is not required in this case).

or b. Female patient of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile. Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges).

Main phase:

Exclusion Criteria:

1. Pregnant or lactating woman where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive pregnancy test (serum pregnancy test to be performed at screening visit and urine pregnancy test to be performed prior to randomization);
2. Run-in compliance to study drug and e-Diary completion < 50% at randomization;
3. History of "high risk" asthma: History of near fatal asthma or hospitalization for asthma in intensive care unit which, in the judgement of the Investigator, may place the subject at undue risk if enrolled in this study;
4. Recent asthma exacerbation: hospitalization, emergency room admission or use of systemic corticosteroids for an asthma exacerbation in the 4 weeks prior to screening visit or during the run-in period;

   Note: Subjects experiencing an exacerbation during the run-in period may be re-screened once, at least 4 weeks after recovery.
5. Non-persistent asthma: exercise-induced, seasonal asthma (as the only asthma-related diagnosis) not requiring daily asthma control medicine;
6. Subjects using systemic corticosteroid medication in the 4 weeks or slow release corticosteroids in the 12 weeks, prior to screening;
7. Asthma requiring use of biologics: Subjects receiving asthma treatment with an injectable biologic drug such as monoclonal antibodies;
8. Respiratory disorders other than asthma: Subjects with known respiratory disorders other than asthma. This can include but is not limited to: diagnosis of COPD as defined by the current guidelines (e.g. GOLD Report), known α1-antitrypsine deficiency, active tuberculosis, bronchiectasis, sarcoidosis, interstitial lung diseases, idiopathic pulmonary fibrosis, and pulmonary hypertension;
9. Lung cancer or history of lung cancer: Subjects with an active diagnosis of lung cancer or a history of lung cancer;
10. Lung resection: Subjects with a history of lung volume resection;
11. Respiratory tract infection: Subjects with respiratory tract infection within 4 weeks prior to screening or during the run-in period; Note: Subjects experiencing a respiratory tract infection during the run-in period may be re-screened once, at least 4 weeks after recovery.
12. Smoking status: Current smoker or ex-smoker with a smoking history of ≥ 10 pack-years (pack-years = the number of cigarette packs per day times the number of years). Ex- smokers must have stopped smoking for ≥1 year (≥ 6 months for e-cigarettes).
13. Cancer or history of cancer (other than lung): Subjects with active cancer or a history of cancer with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localized carcinoma (e.g. basal cell carcinoma, in situ carcinoma of the cervix adequately treated, …) is acceptable;
14. Cardiovascular diseases: Subjects who have clinically significant (CS) cardiovascular condition according to Investigator's judgement, such as but not limited to: congestive heart failure (NYHA class IV), unstable or acute ischemic heart disease in the last year prior to screening, history of sustained and non-sustained cardiac arrhythmias diagnosed in the last 6 months prior to screening (sustained meant lasting more than 30 seconds or ending only with external action, or led to hemodynamic collapse; non-sustained meant > 3 beats < 30 seconds, and or ending spontaneously, and or asymptomatic), high degree impulse conduction blocks (> 2nd degree atrioventricular block type 2),persistent, long standing or paroxysmal atrial fibrillation (AF); Note: Subjects with permanent AF (for at least 6 months prior screening) with a resting ventricular rate < 100/min, controlled with a rate control strategy (i.e. selective β blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) can be considered for enrolment;
15. ECG criteria: Any abnormal and clinically significant 12-lead ECG that in the investigator's opinion would affect efficacy or safety evaluation or place the subjects at risk.
16. ECG QTcF: Male subjects with a Fridericia's corrected QT interval (QTcF) >450 msec and female subjects with a QTcF >470 msec at screening are not eligible (not applicable for subjects with permanent atrial fibrillation and for subjects with pacemaker);
17. Subjects with a medical history or current diagnosis of narrow angle glaucoma, symptomatic prostatic hypertrophy, urinary retention bladder neck obstruction that, in the opinion of the Investigator, would prevent use of anticholinergic agents; Note: Benign prostatic hyperplasia subjects who are stable under treatment can be considered for inclusion.
18. CNS disorders: Subjects with a history of symptoms or significant neurological disease such as but not limited to transient ischemic attack (TIA), stroke, seizure disorder or behavioral disturbances according to the investigator's opinion;
19. Other medical conditions: Subjects with other severe acute or chronic medical or malignancy or psychiatric condition or clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease, that might in the judgment of the Investigator, place the subject at undue risk or potentially compromise the results or interpretation of the study;
20. Other concurrent diseases: Subjects with historical or current evidence of uncontrolled concurrent disease such as but not limited to hyperthyroidism, diabetes mellitus or other endocrine disease; hematological disease; autoimmune disorders (e.g. rheumatoid arthritis, ), gastrointestinal disorders (e..; poorly controlled peptic ulcer, GERD), significant renal and hepatic impairment or other disease or condition that might, in the judgement of the investigator, place the subject at undue risk or potentially compromise the results or interpretation of the study;
21. Liver diseases: Subjects with severe hepatitis, chronic active hepatitis or evidence of uncontrolled chronic liver disease according to the investigator's opinion;
22. Vaccination: Subjects who receive a vaccination within 2 weeks prior to screening or during the run-in;
23. Subjects who have been found to be mentally or legally incapacitate because of an intellectual disability, or subjects who are institutionalized by a government or a judicial order;
24. Contra-indications or Hypersensibiliy to IMPs: Contra-indications to IMPs or hypersensibility to the active substances or to any of the excipients listed in the SmPC of IMPs constitute an exclusion criterion. For warnings, eligibility will be judged by the investigator;
25. Alcohol/drug abuse: Subjects with a history of alcohol or drug abuse within two years prior to the start of the study;
26. Hypersensitivity: Subjects with known intolerance/hypersensitivity or contraindication to treatment with ß2-agonists, ICS, anticholinergics or propellant gases/excipients (as listed in the corresponding SmPCs). For warnings/precaution for use, eligibility will be judged by the investigator;
27. Surgery: Subjects with major surgery in the 3 months prior to screening visit or planned surgery during the trial;
28. Subjects treated with non-potassium sparing diuretics (unless administered as a fixed dose combination [FDC] with a potassium conserving drug or changed to potassium sparing before the screening), nonselective beta blocking drugs, quinidine, quinidine like anti-arrhythmics, or any medication with a corrected QT interval (QTc) prolongation potential or a history of QTc prolongation;
29. Subjects treated with monoamine oxidase inhibitors (MAOIs) and tricyclic anti-depressants;
30. Subjects receiving any therapy that could interfere with the study drugs according to Investigator's opinion;
31. Participation in investigational trial: Subjects who have received an investigational drug within 2 months or six half-lives (whichever is greater) prior to screening visit, or have been previously randomized in this trial, or are currently participating in another clinical trial;
32. Documented coronavirus disease 2019 (COVID-19) diagnosis within 8 weeks prior to screening or its complication which has not resolved within 14 days prior to screening.

Open-label extension phase :

Inclusion criteria:

1. Informed consent: Subject's electronic (preferred option in countries where this is allowed as per local regulations) or written informed consent obtained prior to any study related procedures; Participation in MiSTIC study main phase: Subjects enrolled in MiSTIC main phase, who did not discontinue from the main phase study treatment before Week 26 and with available data to allow classification of asthma control.
2. A willingness and ability:

   * To correctly use the pMDI inhalers;
   * To perform all trial related procedures including technically acceptable pulmonary function tests;
   * To correctly use the e-Diary;
   * To correctly use the technology enabling remote visits and home supervised spirometry assessments (in countries where this is allowed as per local regulations).
3. Treatment compliance during main phase: Subjects with main phase study treatment compliance ≥ 70%
4. Female subjects:

   1. Woman of Childbearing Potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up call or ii. WOCBP with non-fertile male partners (contraception is not required in this case).

      or
   2. Female patient of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile. Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges).

Open-label extension phase:

Exclusion criteria:

1. Pregnant or lactating woman where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive pregnancy test (urine pregnancy test is performed at Visit 6 of the main phase) according to local regulation;
2. Adverse Drug Reactions (ADRs): Subjects who have experienced an ADRs (assessed as possibly related to study drugs by the investigator) during the main phase;
3. Ongoing Serious Adverse Events (SAEs): Subjectswith ongoing SAEs from the main phase at the time of Visit 6 OLE should not be enrolled in the OLE phase unless the investigator considers that the ongoing SAE would not prevent them from safely and effectively participating in the OLE phase;
4. Changes in medical history: Any clinically significant changes in subject's medical history, physical examination (PE)/Vital Signs (VS)/ laboratory analysis; concomitant therapies, documented in the main phase or any new identified disease or condition, that might, in the judgement of the investigator, place the subject at undue risk or potentially compromise the results or interpretation of the study;
5. Changes in study treatments during the main phase or ongoing use of main phase prohibited medications: Any use of biological (monoclonal antibodies e.g. anti-IgE or anti-IgG antibodies) to treat asthma during the main phase or ongoing use of main phase prohibited medications as maintenance treatment for asthma at the time of Visit 6OLE.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Main phase: Proportion of subjects exhibiting No Persistent Airflow Limitation (NPAL) on average over 26 weeks of treatment in the study sub-population with Persistent Airflow Limitation (PAL) status at screening | Over 26 weeks of treatment
  Proportion of subjects exhibiting on average No Persistent Airflow Limitation (NPAL) status over 26 weeks of treatment in the study sub-population meeting Persistent Airflow Limitation (PAL) status at screening. A subject is defined as PAL at screening if post-bronchodilator (salbutamol) FEV1/FVC ratio is < 0.7. A subject is defined as NPAL during the treatment period if the mean of their 2 hour post-dose FEV1/FVC ratio collected during the treatment period is ≥ 0.7
Open-label extension phase: Proportion of subjects that remains or becomes "Adequately Controlled" at the end of the Open-Label extension phase | Over 24 weeks of treatment
  Proportion of subjects that remains or becomes "Adequately Controlled" at the end of the Open-Label extension phase (i.e. Week 50), after the assignment to either MS CHF5993 (BDP/FF/GB 100/6/12.5 pMDI) or HS CHF5993 (BDP/FF/GB 200/6/12.5 pMDI) according to their asthma control status ('Controlled' vs 'Uncontrolled') at the end of MiSTIC main phase (week 26)

SECONDARY OUTCOMES:
Change from baseline in pre-dose FEV1 at Week 26 in the study sub-population meeting PAL criterion at screening | Over 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kostantinos Kostikas, Principal Investigator — Head Respiratory Medicine Department, University Hospital of Ioannina, Greece
Locations (1):
- Simplex Kft, Nyíregyháza, Hungary

IPD SHARING:
Plan to Share IPD: No